CLINICAL TRIAL: NCT02487433
Title: A Phase 1, Randomized, Open Label, Single Dose, 2 Period Crossover Study To Evaluate The Effect Of Food On The Pharmacokinetics Of Tofacitinib Modified Release (mr) 22 Mg Tablets In Healthy Volunteers
Brief Title: A Study To Evaluate The Effect Of Food On The Behavior of Tofacitinib Modified Release 22 Milligram Tablets In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A3921217; 2014-005056-26 (EudraCT Number)
Record Dates: First submitted 2015-04-23; First posted 2015-07-01 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: food effect; pharmacokinetics; healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tofacitinib MR 22 mg Fed (Experimental): Single dose of tofacitinib MR 22 mg administered under fed conditions
  Interventions: Drug: Tofacitinib MR 22 mg (Fed)
- Tofacitinib MR 22 mg Fasted (Experimental): Single dose of tofacitinib MR 22 mg administered under fasted conditions
  Interventions: Drug: Tofacitinib MR 22 mg (Fasted)

INTERVENTIONS:
Drug: Tofacitinib MR 22 mg (Fed) — A single dose of tofacitinib modified release 22 mg tablet after receiving the standard FDA high-fat/high-calorie meal
  Arms: Tofacitinib MR 22 mg Fed
Drug: Tofacitinib MR 22 mg (Fasted) — A single dose of tofacitinib modified release 22 mg tablet after an overnight fast of 10 hours
  Arms: Tofacitinib MR 22 mg Fasted

SUMMARY:
This study will evaluate the drug behavior and safety of a single dose of the 22 milligram tofacitinib (CP-690,550) modified-release formulation in 18 healthy volunteers when taken after eating a high fat meal (the effect of food). This will be compared to the drug behavior and safety of a single dose of the 22 milligram tofacitinib (CP-690,550) modified-release formulation when taken after a 10 hour fast.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers and/or healthy female volunteers of non-childbearing potential who are 18 to 55 years of age;
* Healthy volunteers with no evidence of active or latent or inadequately treated tuberculosis.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease;
* Clinically significant infections within the past 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
AUC inf | 48 hours post dose
  Area under the plasma concentration-time profile from time zero to infinity (AUCinf).
AUC last | 48 hours post dose
  Area under the plasma concentration-time profile from time zero to time of last identifiable quantitation (AUC last).
Cmax | 48 hours post dose
  Maximum observed plasma concentration (Cmax).

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 48 hours post dose
Plasma Decay Half-Life (t 1/2) | 48 hours post dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium